CLINICAL TRIAL: NCT02202551
Title: Open-Label Safety Study of ADS-5102 (Amantadine HCl) Extended Release Capsules for the Treatment of Levodopa Induced Dyskinesia (LID)
Brief Title: Open-Label Safety Study of ADS-5102 in PD Patients With LID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adamas Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADS-AMT-PD302
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-08

CONDITIONS: Dyskinesia; Levodopa Induced Dyskinesia (LID); Parkinson's Disease (PD)
Keywords: Levodopa Induced Dyskinesia; LID; Parkinsonism; Parkinson's Disease
MeSH Terms: conditions — Dyskinesias; Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADS-5102 (Experimental): amantadine HCl extended release
  Interventions: Drug: ADS-5102

INTERVENTIONS:
Drug: ADS-5102
  Other Names: amantadine HCl extended release

SUMMARY:
This is a 105-week open-label study to evaluate the safety and tolerability of ADS-5102 oral capsules, an extended release formulation of amantadine, in Parkinson's Disease (PD) patients with Levodopa Induced Dyskinesia (LID).

DETAILED DESCRIPTION:
Participation in this study was offered to subjects who were described by one of the following 3 groups:

* Group 1: Subjects who completed an Adamas efficacy study evaluating ADS-5102 in LID and chose to immediately transition into the current study without a time gap; this group was subdivided into Group 1A, consisting of subjects who received ADS-5102 in the previous Adamas efficacy study, and Group 1P, consisting of subjects who received placebo in the previous Adamas efficacy study
* Group 2: Subjects who completed a previous Adamas efficacy study evaluating ADS-5102 in LID and entered the current study with a time gap
* Group 3: Subjects who would have been deemed ineligible for participation in a previous Adamas efficacy study due to having undergone DBS

Consented subjects who completed Screening (Visit 1) and met study eligibility criteria were to have a Baseline Visit and receive study drug. During Week 1, subjects took 170 mg of ADS-5102 (1 capsule) daily at bedtime. For Week 2, the dose was increased to 340 mg (2 capsules) daily at bedtime; this dose was to continue through Week 100. During the final week (Week 101) of the study, the ADS-5102 dose was reduced to 170 mg (1 capsule) daily at bedtime. Subjects were enrolled into the study at Visit 2 (Baseline/Week 0) and were to return to the clinic after 4, 8, 16, 28, 40, 52, 64, 76, 88, and 100 weeks of study drug dosing. Subjects were to receive a telephone reminder at the end of Week 1 to increase their dose during Week 2. At the Week 100 Visit, subjects were instructed to reduce their dose to 1 capsule daily at bedtime for 1 week. The amount of available, unused drug was assessed during the Week 100 Visit; subjects were given an additional bottle of study drug, if needed, to complete the 1 week of reduced dosing.

Efficacy, as measured with the MDS-UPDRS, was to be evaluated at all study visits, beginning with the Screening Visit, and excluding the Baseline and Week 4 Visits. A Safety Follow-up Visit was to occur approximately 2 weeks following the completion of treatment. AEs were recorded beginning with the first dose of study drug and continued through the Safety Follow-up Visit. Concomitant medications were recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed a current IRB/REB/IEC-approved informed consent form
* Completed all study visits in previous Adamas efficacy study or were ineligible for participation in previous Adamas studies due to having undergone prior deep brain stimulation.
* Parkinson's disease, per UK Parkinson's Disease Society (UKPDS) Brain Bank Clinical Diagnostic Criteria
* On a stable regimen of antiparkinson's medications at least 30 days prior to screening, including a levodopa preparation administered not less than three times daily.
* History of peak dose dyskinesia that might benefit from specific dyskinesia treatment in the judgment of the subject and clinical investigator

Exclusion Criteria:

* Discontinued ADS-5102 in previous Adamas efficacy study due to intolerable or unacceptable AEs considered to be related to ADS-5102
* History of neurosurgical intervention related to Parkinson's disease, with the exception of deep brain stimulation
* History of seizures since completion of participation in previous Adamas studies or within 2 years
* History of stroke or TIA since completion of participation in previous Adamas studies or within 2 years
* History of cancer since completion of participation in previous Adamas studies or within 2 years, with the following exceptions: adequately treated non-melanomatous skin cancers, localized bladder cancer, non-metastatic prostate cancer or in situ cervical cancer
* Presence of cognitive impairment, as evidenced by a Mini-Mental Status Examination (MMSE) score of less than 24 during screening
* If female is pregnant or lactating
* If a sexually active female, is not surgically sterile or at least 2 years post-menopausal, or does not agree to utilize an effective method of contraception from screening through at least 4 weeks after the completion of study treatment.
* Treatment with an investigational drug (other than ADS-5102) or device within 30 days prior to screening
* Treatment with an investigational biologic within 6 months prior to screening
* Current or planned participation in another interventional clinical trial

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2014-07; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Director, Study Director — Adamas Pharmaceuticals, Inc.
Locations (76):
- United States (49):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Sun City, Arizona
  - Fountain Valley, California
  - Pasadena, California
  - Reseda, California
  - Sacramento, California
  - Sunnyvale, California
  - Torrance, California
  - Ventura, California
  - Aurora, Colorado
  - Manchester, Connecticut
  - Boca Raton, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Naples, Florida
  - Port Charlotte, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - Weston, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Baltimore, Maryland
  - Elkridge, Maryland
  - Boston, Massachusetts
  - Bingham Farms, Michigan
  - West Bloomfield, Michigan
  - Golden Valley, Minnesota
  - St Louis, Missouri
  - Albany, New York
  - Commack, New York
  - New York, New York
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - Roanoke, Virginia
  - Kirkland, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Austria (2):
  - Innsbruck
  - Vienna
- Canada (3):
  - Edmonton, Alberta
  - Toronto, Ontario
  - Regina, Saskatchewan
- France (11):
  - Bordeaux
  - Bron
  - Clermont-Ferrand
  - Lille
  - Marseille
  - Montpellier
  - Poitiers
  - Rennes
  - Rouen
  - Strasbourg
  - Toulouse
- Germany (10):
  - München, Bavaria
  - Beelitz-Heilstätten, Brandenburg
  - Göttingen, Lower Saxony
  - Leipzig, Saxony
  - Gera, Thuringia
  - Stadtroda, Thuringia
  - Berlin
  - Hamburg
  - Kassel
  - Marburg
- Barcelona, Spain

REFERENCES:
- [Background] Aoki FY, Sitar DS. Clinical pharmacokinetics of amantadine hydrochloride. Clin Pharmacokinet. 1988 Jan;14(1):35-51. doi: 10.2165/00003088-198814010-00003. PMID 3280212
- [Background] Colosimo C, Martinez-Martin P, Fabbrini G, Hauser RA, Merello M, Miyasaki J, Poewe W, Sampaio C, Rascol O, Stebbins GT, Schrag A, Goetz CG. Task force report on scales to assess dyskinesia in Parkinson's disease: critique and recommendations. Mov Disord. 2010 Jul 15;25(9):1131-42. doi: 10.1002/mds.23072. PMID 20310033
- [Background] da Silva-Junior FP, Braga-Neto P, Sueli Monte F, de Bruin VM. Amantadine reduces the duration of levodopa-induced dyskinesia: a randomized, double-blind, placebo-controlled study. Parkinsonism Relat Disord. 2005 Nov;11(7):449-52. doi: 10.1016/j.parkreldis.2005.05.008. Epub 2005 Sep 9. PMID 16154788
- [Background] Dallos V, Heathfield K, Stone P, Allen FA. Use of amantadine in Parkinson's disease. Results of a double-blind trial. Br Med J. 1970 Oct 3;4(5726):24-6. doi: 10.1136/bmj.4.5726.24. PMID 4919119
- [Background] Del Sorbo F, Albanese A. Levodopa-induced dyskinesias and their management. J Neurol. 2008 Aug;255 Suppl 4:32-41. doi: 10.1007/s00415-008-4006-5. PMID 18821084
- [Background] Encarnacion EV, Hauser RA. Levodopa-induced dyskinesias in Parkinson's disease: etiology, impact on quality of life, and treatments. Eur Neurol. 2008;60(2):57-66. doi: 10.1159/000131893. Epub 2008 May 15. PMID 18480609
- [Background] Factor SA, Molho ES. Transient benefit of amantadine in Parkinson's disease: the facts about the myth. Mov Disord. 1999 May;14(3):515-7. doi: 10.1002/1531-8257(199905)14:33.0.co;2-z. No abstract available. PMID 10348482
- [Background] Goetz CG, Nutt JG, Stebbins GT. The Unified Dyskinesia Rating Scale: presentation and clinimetric profile. Mov Disord. 2008 Dec 15;23(16):2398-403. doi: 10.1002/mds.22341. PMID 19025759
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Goetz CG, Stebbins GT, Chung KA, Hauser RA, Miyasaki JM, Nicholas AP, Poewe W, Seppi K, Rascol O, Stacy MA, Nutt JG, Tanner CM, Urkowitz A, Jaglin JA, Ge S. Which dyskinesia scale best detects treatment response? Mov Disord. 2013 Mar;28(3):341-6. doi: 10.1002/mds.25321. Epub 2013 Feb 6. PMID 23390076
- [Background] Hayden FG, Gwaltney JM Jr, Van de Castle RL, Adams KF, Giordani B. Comparative toxicity of amantadine hydrochloride and rimantadine hydrochloride in healthy adults. Antimicrob Agents Chemother. 1981 Feb;19(2):226-33. doi: 10.1128/AAC.19.2.226. PMID 7347558
- [Background] Jackson G, Stanley E, Lee Muldoon R. Chemoprophylaxis of viral respiratory diseases. Bulletin Pan Am Health Org. 1967; 147: 595-603.
- [Background] Luginger E, Wenning GK, Bosch S, Poewe W. Beneficial effects of amantadine on L-dopa-induced dyskinesias in Parkinson's disease. Mov Disord. 2000 Sep;15(5):873-8. doi: 10.1002/1531-8257(200009)15:53.0.co;2-i. PMID 11009193
- [Background] Ory-Magne F, Corvol JC, Azulay JP, Bonnet AM, Brefel-Courbon C, Damier P, Dellapina E, Destee A, Durif F, Galitzky M, Lebouvier T, Meissner W, Thalamas C, Tison F, Salis A, Sommet A, Viallet F, Vidailhet M, Rascol O; NS-Park CIC Network. Withdrawing amantadine in dyskinetic patients with Parkinson disease: the AMANDYSK trial. Neurology. 2014 Jan 28;82(4):300-7. doi: 10.1212/WNL.0000000000000050. Epub 2013 Dec 26. PMID 24371304
- [Background] Paci C, Thomas A, Onofrj M. Amantadine for dyskinesia in patients affected by severe Parkinson's disease. Neurol Sci. 2001 Feb;22(1):75-6. doi: 10.1007/s100720170054. PMID 11487209
- [Background] Parkes JD, Zilkha KJ, Marsden P, Baxter RC, Knill-Jones RP. Amantadine dosage in treatment of Parkinson's disease. Lancet. 1970 May 30;1(7657):1130-3. doi: 10.1016/s0140-6736(70)91211-0. No abstract available. PMID 4192093
- [Background] Sawada H, Oeda T, Kuno S, Nomoto M, Yamamoto K, Yamamoto M, Hisanaga K, Kawamura T; Amantadine Study Group. Amantadine for dyskinesias in Parkinson's disease: a randomized controlled trial. PLoS One. 2010 Dec 31;5(12):e15298. doi: 10.1371/journal.pone.0015298. PMID 21217832
- [Background] Schrag A, Quinn N. Dyskinesias and motor fluctuations in Parkinson's disease. A community-based study. Brain. 2000 Nov;123 ( Pt 11):2297-305. doi: 10.1093/brain/123.11.2297. PMID 11050029
- [Background] Schwab RS, Poskanzer DC, England AC Jr, Young RR. Amantadine in Parkinson's disease. Review of more than two years' experience. JAMA. 1972 Nov 13;222(7):792-5. doi: 10.1001/jama.222.7.792. No abstract available. PMID 4677928
- [Background] Snow BJ, Macdonald L, Mcauley D, Wallis W. The effect of amantadine on levodopa-induced dyskinesias in Parkinson's disease: a double-blind, placebo-controlled study. Clin Neuropharmacol. 2000 Mar-Apr;23(2):82-5. doi: 10.1097/00002826-200003000-00004. PMID 10803797
- [Background] Spencer TJ, Biederman J, Ciccone PE, Madras BK, Dougherty DD, Bonab AA, Livni E, Parasrampuria DA, Fischman AJ. PET study examining pharmacokinetics, detection and likeability, and dopamine transporter receptor occupancy of short- and long-acting oral methylphenidate. Am J Psychiatry. 2006 Mar;163(3):387-95. doi: 10.1176/appi.ajp.163.3.387. PMID 16513858
- [Background] Swanson JM, Volkow ND. Pharmacokinetic and pharmacodynamic properties of stimulants: implications for the design of new treatments for ADHD. Behav Brain Res. 2002 Mar 10;130(1-2):73-8. doi: 10.1016/s0166-4328(01)00433-8. PMID 11864720
- [Background] Thomas A, Iacono D, Luciano AL, Armellino K, Di Iorio A, Onofrj M. Duration of amantadine benefit on dyskinesia of severe Parkinson's disease. J Neurol Neurosurg Psychiatry. 2004 Jan;75(1):141-3. PMID 14707325
- [Background] Tyrrell DA, Bynoe ML, Hoorn B. Studies on the antiviral activity of 1-adamantanamine. Br J Exp Pathol. 1965 Aug;46(4):370-5. No abstract available. PMID 5317962
- [Background] Verhagen Metman L, Del Dotto P, van den Munckhof P, Fang J, Mouradian MM, Chase TN. Amantadine as treatment for dyskinesias and motor fluctuations in Parkinson's disease. Neurology. 1998 May;50(5):1323-6. doi: 10.1212/wnl.50.5.1323. PMID 9595981
- [Background] Metman LV, Del Dotto P, LePoole K, Konitsiotis S, Fang J, Chase TN. Amantadine for levodopa-induced dyskinesias: a 1-year follow-up study. Arch Neurol. 1999 Nov;56(11):1383-6. doi: 10.1001/archneur.56.11.1383. PMID 10555659
- [Background] Volkow ND, Wang GJ, Fowler JS, Gatley SJ, Logan J, Ding YS, Hitzemann R, Pappas N. Dopamine transporter occupancies in the human brain induced by therapeutic doses of oral methylphenidate. Am J Psychiatry. 1998 Oct;155(10):1325-31. doi: 10.1176/ajp.155.10.1325. PMID 9766762
- [Background] Wolf E, Seppi K, Katzenschlager R, Hochschorner G, Ransmayr G, Schwingenschuh P, Ott E, Kloiber I, Haubenberger D, Auff E, Poewe W. Long-term antidyskinetic efficacy of amantadine in Parkinson's disease. Mov Disord. 2010 Jul 30;25(10):1357-63. doi: 10.1002/mds.23034. PMID 20198649
- [Background] Wright Willis A, Evanoff BA, Lian M, Criswell SR, Racette BA. Geographic and ethnic variation in Parkinson disease: a population-based study of US Medicare beneficiaries. Neuroepidemiology. 2010;34(3):143-51. doi: 10.1159/000275491. Epub 2010 Jan 15. PMID 20090375
- [Derived] Hauser RA, Pahwa R, Tanner CM, Oertel W, Isaacson SH, Johnson R, Felt L, Stempien MJ. ADS-5102 (Amantadine) Extended-Release Capsules for Levodopa-Induced Dyskinesia in Parkinson's Disease (EASE LID 2 Study): Interim Results of an Open-Label Safety Study. J Parkinsons Dis. 2017;7(3):511-522. doi: 10.3233/JPD-171134. PMID 28777755

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1a: Subjects completed previous LID study and enrolled in ADS-AMT-PD302 study immediately. Subjects in Group 1A received ADS-5102 in the prior study.
- Group 1P: Subjects completed previous LID study and enrolled in ADS-AMT-PD302 study immediately. Subjects in Group 1P received placebo in the prior study
- Group 2: Subjects in Group 2 completed previous LID study, enrolled ADS-AMT-PD302 after a time gap.
- Group 3: Subjects were not in a previous Adamas LID study and had prior DBS (deep brain stimulation)
Period: Overall Study
Arm/Group | Group 1a | Group 1P | Group 2 | Group 3
Started | 60 | 78 | 24 | 61
Completed | 35 | 41 | 14 | 39
Not Completed | 25 | 37 | 10 | 22
Not completed — Adverse Event | 8 | 19 | 5 | 9
Not completed — Death | 3 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Needed to take excluded medication | 0 | 2 | 0 | 1
Not completed — Subject moved away | 0 | 1 | 0 | 0
Not completed — DBS surgery | 3 | 0 | 0 | 0
Not completed — Dyskinesia upon taper | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Site closure | 3 | 0 | 0 | 1
Not completed — Unable to complete visits per protocol | 1 | 0 | 0 | 0
Not completed — Worsening Dyskinesia | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Sponsor's decision | 2 | 0 | 0 | 0
Not completed — Subject unwilling to proceed | 1 | 5 | 3 | 5
Not completed — Subject consent withdrawn | 0 | 3 | 1 | 2
Not completed — eGFR<50mL/min/m2 | 2 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1a | Group 1P | Group 2 | Group 3 | Total
Number analyzed (Participants) | 60 | 78 | 24 | 61 | 223
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 30 | 12 | 39 | 109
  >=65 years | 32 | 48 | 12 | 22 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.81) | 65.9 (8.80) | 64.4 (7.81) | 60.2 (9.20) | 63.7 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 33 | 13 | 20 | 92
  Male | 34 | 45 | 11 | 41 | 131
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 57 | 74 | 23 | 54 | 208
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 2 | 5
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.86 (25.42) | 25.72 (24.63) | 25.26 (23.24) | 27.29 (4.891) | 26.14 (5.220)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 88.7 (24.31) | 92.2 (19.64) | 96.3 (20.54) | 92.1 (19.95) | 91.6 (21.16)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reported AEs and Safety-Related Study Drug Discontinuations
Description: The primary objective of the study was to evaluate the safety and tolerability of ADS-5102 oral capsules, an extended release (ER) formulation of amantadine, administered at a dose of 340 mg once daily at bedtime for the treatment of levodopa-induced dyskinesia (LID) in subjects with Parkinson's disease (PD).
Time Frame: Up to 101 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a | Group 1P | Group 2 | Group 3
Number analyzed (Participants) | 60 | 78 | 24 | 61
Participants
  AE | 57 | 70 | 23 | 55
  Study drug-related AE | 31 | 45 | 16 | 32
  SAEs | 16 | 21 | 6 | 17
  Permanent discontinuation due to AE | 12 | 21 | 6 | 10
  Permanent discontinuation due to drug-related AE | 4 | 15 | 4 | 8
  Mild AEs | 12 | 13 | 3 | 11
  Moderate AEs | 25 | 36 | 13 | 26
  Mild drug-related AE | 16 | 15 | 3 | 5
  Moderate drug-related AE | 12 | 23 | 12 | 22
  Severe drug-related AE | 3 | 7 | 1 | 5

2. Secondary Outcome: Change From Baseline in Movement Disorder's Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) (Parts I-III Combined Scores)
Description: To evaluate clinical progression of PD as assessed by the MDS-UPDRS, combined score, Parts I, II, and III.
  Part I - non-motor experiences of daily living; Part II - motor experiences of daily living; Part III - motor examination. Parts I and II each contain 13 questions measured on a 5-point scale (0-4). Part III contains 18 objective rater assessments of the motor signs of PD measured on a 5-point scale (0-4).
  Total range for combined score (Part I-III) is = 0-176. Generally for MDS-UPDRS scores and sub-scores, the lower the score, the better.
  Parts I, II, and III are summed to make the total score.
Time Frame: Up to 101 weeks. MDS-UPDRS was performed at the following visits: Screening, Week 8, Week 16, Week 28, Week 40, Week 52, Week 64, Week 76, Week 88, Week 100 (or ET).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ADS-5102 1A: Consisting of subjects who received ADS-5102 in the previous Adamas efficacy study
- ADS-5102 Group 1P: Consisting of subjects who received placebo in the previous Adamas efficacy study
- ADS-5102 Group 2: Subjects who completed a previous Adamas efficacy study evaluating ADS-5102 in LID and entered the current study with a time gap
- ADS-5102 Group 3: Subjects who would have been deemed ineligible for participation in a previous Adamas efficacy study due to having undergone DBS
Arm/Group | ADS-5102 1A | ADS-5102 Group 1P | ADS-5102 Group 2 | ADS-5102 Group 3
Number analyzed (Participants) | 60 | 77 | 24 | 60
units on a scale
  Baseline | 41.8 (18.43) | 45.6 (19.24) | 52.8 (23.06) | 52.4 (16.55)
  Change from Baseline at Week 8 | 1.2 (10.03) | -2.8 (14.11) | 0.8 (12.00) | -5.3 (10.74)
  Change from Baseline at Week 16 | 1.6 (13.41) | -1.4 (16.22) | 5.7 (15.53) | -5.2 (11.33)
  Change from Baseline at Week 28 | 4.8 (10.04) | 1.5 (12.49) | 6.5 (14.18) | -5.3 (12.99)
  Change from Baseline at Week 40 | 7.5 (15.43) | -0.4 (15.20) | 1.6 (18.29) | -4.8 (12.49)
  Change from Baseline at Week 52 | 13.2 (16.78) | 2.6 (14.57) | 6.1 (18.34) | -4.6 (15.60)
  Change from Baseline at Week 64 | 8.8 (14.83) | 2.6 (14.57) | 6.1 (18.34) | -4.6 (15.60)
  Change from Baseline at Week 76 | 11.7 (19.58) | 7.3 (19.18) | 9.4 (19.10) | -4.9 (13.83)
  Change from Baseline at Week 88 | 11.3 (16.65) | 3.7 (13.80) | 6.4 (22.65) | 0.9 (16.18)
  Change from Baseline at Week 100 | 11.4 (15.66) | 3.7 (15.29) | 6.5 (16.46) | 4.1 (17.48)

3. Secondary Outcome: Change From Baseline in Movement Disorder's Society - Unified Parkinson's Disease Rating Scale MDS-UPDRS (Part IV - Motor Complications)
Description: This component (Questions 4.1 - 4.6) includes time spent with dyskinesia, functional impact of dyskinesia, time spent in OFF state, functional impact of fluctuations, complexity of motor fluctuations, painful OFF-state dystonia. Questions 4.1-4.6 are summed to make the Part IV score.
  Generally for MDS-UPDRS scores and sub-scores, the lower the score, the better. Total range for Part IV is = 0-24
Time Frame: 100 Weeks. MDS-UPDRS was performed at the following visits: Screening, Week 8, Week 16, Week 28, Week 40, Week 52, Week 64, Week 76, Week 88, Week 100 (or ET).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1a | Group 1P | Group 2 | Group 3
Number analyzed (Participants) | 60 | 77 | 24 | 60
units on a scale
  Baseline | 6.5 (3.38) | 9.6 (3.07) | 9.8 (3.92) | 10.4 (2.77)
  Change in Baseline from Week 8 | -0.2 (3.21) | -3.4 (3.27) | -3.6 (4.16) | -4.0 (4.20)
  Change in Baseline from Week 16 | -0.8 (3.61) | -3.2 (3.61) | -1.1 (5.03) | -3.9 (3.68)
  Change from Baseline at Week 28 | -0.3 (3.61) | -3.3 (3.12) | -1.4 (3.84) | -4.4 (3.79)
  Change from Baseline at Week 40 | 0.0 (3.95) | -2.8 (3.39) | -2.9 (4.81) | -4.7 (4.06)
  Change from Baseline at Week 52 | 0.2 (3.64) | -2.9 (3.56) | -2.5 (4.40) | -3.6 (3.62)
  Change from Baseline at Week 64 | 0.4 (3.82) | -3.3 (3.42) | -1.9 (4.32) | -2.5 (4.22)
  Change from Baseline at Week 76 | 0.9 (4.20) | -2.9 (3.67) | -2.7 (3.90) | -3.7 (3.68)
  Change from Baseline at Week 88 | 0.4 (3.77) | -2.8 (3.60) | -3.7 (4.69) | -4.3 (3.55)
  Change from Baseline at Week 100 | 0.4 (3.28) | -2.4 (4.19) | -3.6 (3.66) | -3.6 (3.94)

ADVERSE EVENTS:
Time Frame: 100 weeks
Description: Safety was assessed through adverse events (AEs), physical examinations, vital signs, and laboratory parameters (hematology, serum chemistry, urinalysis, and pregnancy testing, if appropriate).
Arm/Group | Group 1a | Group 1P | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 4/60 | 2/78 | 2/24 | 1/61
Serious Adverse Events (participants affected / at risk) | 16/60 | 21/78 | 6/24 | 17/61
Other Adverse Events (participants affected / at risk) | 47/60 | 61/78 | 21/24 | 45/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1a (N=60) | Group 1P (N=78) | Group 2 (N=24) | Group 3 (N=61)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Acute colitis
Ostenecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Avascular necrosis of the right patella
Arthritis bacteria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Septic right knee requiring right total nee arthroplasty
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-St-Elevation mycardial infarction
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Supraventricular tachycardia
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Sigmoid, volvulus
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Worsening right knee degenerative disease
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Oglive Syndrome
Clostridium difficile sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — C. diff sepsis
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Left knee laceration
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Slow transit constipation
Psychiatric disorder (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) — Psychosis
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Septic shock
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Encephalopathy
Lymphoadenopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Lymphoadenopathy
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Right distal radius fracture
Adenocarcinoma of the colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Adenocarcinoma of the ascending colon (right)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Acute confusional syndrome
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Pseudomona aeruginosa sepsis
Neuroleptic malignant syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Malignant neuroleptic syndrome
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Intestinal oclusion
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Ribs fracture
Parkinson's disease (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2) — Worsening of Parkinson's disease
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Shoulder luxation
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Cardiac arrest
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Comminuted intertrichanteric right hip fracture
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Fractured right ankle
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Persistent urinary tract infection
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Rhabdomyolysis
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Cardiac chest pain (etiology unknown)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Adverse drug reaction to melatonin and stool softner
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Heart attack
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Left hip fracture
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Left intertrochanteric femur fracture
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Cardiac arrhythmia
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Intestinal obstruction
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Attempted suicide
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Respiratory arrest
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Angina pectoris due to coronary vascular disease
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Paraesthesia
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Traumatic serial rib fractures
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hemothorax
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Acetabulum fracture right
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Fractured pelvis
On and Off Phenomenon (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Worsening motor fluctuations related to PD
Confusion postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Confusion after hip prothesis surgery
Restless leg syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Worsening of restless leg syndrome
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Abdominal pain (obstipation)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Left wrist fracture
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pneumonia
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — MRSA bacteremia, presumably due to infected hardware
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Respiratory distress secondary to pneumonia
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Worsening of right knee pain
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Worsening benign prostatic hypertrophy
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Cellulitis - right leg
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Altered mental status
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Death due to natural causes
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Sepsis
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Right tibial fracture - motor vehicle accident
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Altered mental state, confusion (occurred 30 days after the last dose)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Broken ankle (left)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Worsening anxiety
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Suicidal ideation with intent for self harm
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Dysfunction of deep brain stimulation device with increased disposition to fall
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Benign paroxysmal positional vertigo
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Craniocerebral injury
Hypokinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hypokinesis
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Intercostal neuralgia
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Forearm fracture left
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hypertensive crisis
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Tongue swelling due to allergic reaction
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Thrombosis of the vena saphena magna in the thigh and lower leg left side
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Semi-myocardial infarction
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Parkinsonism aggravation
Hypertensive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hypertensive cardiomyopathy
Abasia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unable to walk
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Anterior myocardial infarction with acute pulmonary edema
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Left knee join effusion
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Acute psychiatric disorder (maniac manifestation)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Worsening of dyskinesia (reassessment about alternative therapeutic)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Epigastralgia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1a (N=60) | Group 1P (N=78) | Group 2 (N=24) | Group 3 (N=61)
Fall (Injury, poisoning and procedural complications) | 13 | 29 | 8 | 23 — Fall
Hallucination (pooled) (Psychiatric disorders) | 15 | 24 | 5 | 10 — Hallucination (Pooled = combines all Preferred terms that contain the term "Hallucination."
Hallucination, visual (Psychiatric disorders) | 14 | 24 | 4 | 10
Edema peripheral (General disorders) | 10 | 12 | 2 | 12
Constipation (Gastrointestinal disorders) | 9 | 12 | 6 | 3
Urinary tract infection (Infections and infestations) | 7 | 8 | 3 | 5
Dizziness (Nervous system disorders) | 4 | 10 | 5 | 3
Nausea (Gastrointestinal disorders) | 7 | 8 | 6 | 1
Insomnia (Psychiatric disorders) | 8 | 5 | 4 | 4
Livedo reticularis (Skin and subcutaneous tissue disorders) | 6 | 5 | 3 | 6
On and off phenomenon (Nervous system disorders) | 7 | 4 | 4 | 3 — These events were worsening of disease over the duration of the study
Dry mouth (Gastrointestinal disorders) | 4 | 6 | 4 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 2 | 4
Depression (Psychiatric disorders) | 4 | 5 | 2 | 4
Parkinson's disease (Nervous system disorders) | 3 | 5 | 1 | 6 — Worsening of Parkinson's disease
Anxiety (Psychiatric disorders) | 3 | 6 | 1 | 4
Abnormal dreams (Psychiatric disorders) | 5 | 4 | 2 | 2
Nasopharyngitis (Infections and infestations) | 4 | 4 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 1 | 1
Hypertension (Cardiac disorders) | 2 | 6 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT02202551/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT02202551/SAP_001.pdf